CLINICAL TRIAL: NCT06058624
Title: Assessing the Efficacy of an Acceptance-Based Digital Intervention to Improve Functioning for Veterans With Chronic Pain
Brief Title: Assessing the Efficacy of an Acceptance-Based Digital Intervention for Veterans With Chronic Pain
Acronym: VACT-CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: North Texas Veterans Healthcare System (U.S. Federal Agency); VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4804-R; RX004804-01 (Other Grant/Funding Number: VA Office of Research and Development (ORD))
Record Dates: First submitted 2023-09-18; First posted 2023-09-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Internet-Based Intervention; Psychosocial Intervention; Acceptance and Commitment Therapy; Quality of Life; Veterans
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Two arm, randomized clinical trial comparing two online pain self-management interventions: Veteran ACT for Chronic Pain and Online Pain School. Both interventions are matched for attention and time, with 7 modules (each about 15 - 20 minutes) received over 7 weeks.
Who Masked: Outcomes Assessor
Masking Description: The research staff collecting trial outcome data will not be informed of the participant's group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veteran ACT for Chronic Pain (VACT-CP) (Experimental): Participants will complete seven modules (each approximately 15 minutes) over seven weeks. The purpose of VACT-CP is to assist with at home therapeutic and behavioral self-management of chronic pain, based on the principles of acceptance and commitment therapy. Following the end of treatment (7 weeks), participants will complete post-treatment surveys at Week 7, Month 3, and Month 6 to provide feedback and information regarding 1) the intervention and 2) the potential impact of the intervention on functioning, quality of life, and other mental and physical health factors.
  Interventions: Behavioral: Veteran ACT for Chronic Pain (VACT-CP)
- Online Pain School (Active Comparator): Participants will complete seven modules (each approximately 15 minutes) over seven weeks. Online Pain School is designed to balance for time participating in the intervention, and is also an active online attention control. The goal of this program will be to provide Veterans with more tools and options for pain management, and the online format will allow us to monitor website use/dose. Following the end of treatment (7 weeks), participants will complete post-treatment surveys at Week 7, Month 3, and Month 6 to provide feedback and information regarding 1) the intervention and 2) the potential impact of the intervention on functioning, quality of life, and other mental and physical health factors.
  Interventions: Behavioral: Online Pain School

INTERVENTIONS:
Behavioral: Veteran ACT for Chronic Pain (VACT-CP) — Participants receive 7 online modules, provided as weekly sessions that feature Coach Anne as a virtual, animated treatment guide. All content is presented interactively, through text-based conversations with Coach Anne. Veterans will hear what Coach Anne "says" and respond to her using text-based dialogue options that will trigger different responses from Coach Anne as the conversation progresses, to allow the system to responsively interact in a personalized manner with the Veteran. Veterans will also be presented with videos (e.g., Veteran narratives, metaphors), in-module assessments (e.g., values assessments), and interactive opportunities for goal setting.
  Arms: Veteran ACT for Chronic Pain (VACT-CP)
Behavioral: Online Pain School — Participants will receive 7 modules (15 to 20 minutes each) of content based on a common non-ACT based VA treatment option, Pain School. The adaptation used for this study, "Online Pain School", will support Veterans' self-management of their chronic pain by providing informational videos on chronic pain and its health impacts, short behavioral exercises to help with pain management, and psychoeducation on different wellness techniques for their "pain management toolbox."
  Arms: Online Pain School

SUMMARY:
Pain has been identified as among the most frequent presenting medical complaints, in particular within primary care for Veterans. There are few areas of daily living and functioning that pain intensity does not impact, with reported pain intensity related to difficulties in social situations and changes in activities of daily life, sleep, and appetite. Therapeutic interventions such as Acceptance and Commitment Therapy for Chronic Pain (ACT-CP) that target issues related to the cognitions and emotional concerns related to chronic pain have been well-documented for reduction of associated psychiatric symptoms and modest pain relief. At the same time, online programming can improve the ability of pain psychoeducation programs and ACT-CP to reach patients. The proposed project will compare online Veteran ACT for Chronic Pain (VACT-CP) compared to another pain program, Online Pain School, to evaluate how they assist Veterans with chronic pain to improve their functioning, pain management, and quality of life.

DETAILED DESCRIPTION:
Chronic pain is a serious concern that disproportionately affects Veterans compared to the general public; Veterans are diagnosed with CP at particularly high rates (47 - 56%) with a 40% greater rate of severe pain than non-Veterans. Veterans with chronic pain face numerous negative functional outcomes, including decreased ability to complete daily work activities, less social support from and closeness with family members, increased chronic health conditions (e.g., cancer, heart disease), and higher mortality compared to Veterans without chronic pain. Unfortunately, the use of medication for long-term pain treatment, though often utilized, has both limited efficacy and potentially harmful outcomes. Given these concerns, there is an urgent need for innovative and integrative approaches for non-medical pain self-management management. Despite the critical importance of effective pain self-management programs, many Veterans with chronic pain do not engage in pain self-management programs available through the VA. There are numerous reasons for this, including perceived time and transportation concerns and pain-related barriers to attending in-person care options. To improve Veterans' quality of life and it is important to develop and evaluate innovative, accessible, evidence-based interventions for managing pain that can be easily accessed where healthcare happens most - within the home.

One approach with over twenty years of efficacious treatment for chronic pain is Acceptance and Commitment Therapy for Chronic Pain (ACT-CP). ACT is a well-established and VA-approved approach to chronic pain management, and focuses on committing to behavior change that reflects personal values, leading to significant improvement in life functioning. Though provided at many VA hospitals, clinician-delivered ACT for chronic pain has not had a nationwide rollout and is not available at all VA pain clinics. Additionally, many Veterans with chronic pain do not access one-on-one therapeutic treatment due to transportation and time issues. Thankfully, for adults with chronic pain outside of the VA, technology-delivered ACT has been found to be acceptable, useful, and efficacious in delivering pain treatment. However, although research suggests it could help with at-home pain management, no ACT for chronic pain online treatment exists specifically for Veterans and their particular care needs.

To address this treatment option gap, the research team created an online Veteran ACT for chronic pain (VACT-CP) during the PI's Rehabilitation R&D CDA-2 project. VACT-CP is guided by an interactive virtual coach (Coach Anne) to help address pain-related distress and functional difficulties of chronic pain (e.g., avoidance, reactivity) over seven weeks of treatment. Preliminary findings suggest that VACT-CP is highly usable, perceived as helpful, and can help Veterans increase their pain acceptance and pain management. The primary outcomes for this project will be to complete a three-site, fully-powered efficacy trial comparing VACT-CP to an active online control condition (total n = 200) to investigate whether VACT-CP can improve pain-related functioning and quality of life. In addition, the investigators will analyze data from the VACT-CP group to assess whether the hypothesized mechanism of change (psychological flexibility) mediates the impact of pain severity on pain-related functioning.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of non-cancer chronic pain, defined by:

  * 1a at least one pain-related diagnosis indicated by an ICD-9 or -10 code related to either Musculoskeletal pain or Joint Problems/Osteoarthritis
  * 1b. minimum Grade 1 or 2 on the Graded Chronic Pain Scale
* Has a computer and working, high-speed wireless internet connection at home
* Competent to provide written informed consent

Exclusion Criteria:

* Any current or lifetime DSM-5 psychotic disorder
* Current or recent (within 1 month of study entry) DSM-5 substance use disorder
* Current use of any other chronic pain-related psychological treatment
* Clinically significant suicidality within the past year
* Any cognitive or physical impairment that would interfere with study participation of using a computer and providing feedback

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory Change | Week 7, 3-Month Follow-Up, 6 Month Follow-Up
  The Brief Pain Inventory is a widely-used assessment of both pain-relevant functioning and pain severity which is sensitive to change across numerous treatment studies. The pain severity index (BPI-Pain Severity) consists of four items used to assess pain severity and the pain interference scale (BPI-Interference) consists of 7 items that assess the degree of pain interference with functioning across 7 areas: general activity, mood, walking ability, normal work, relationships, sleep; and enjoyment in life. Items are rated on a 0-10 (0 = no pain/no interference and 10 = most pain/most interference).
Veteran's RAND 36 Item Health Survey (VR-36) Change | Week 7, 3-Month Follow-Up, 6 Month Follow-Up
  The Veteran's RAND 36 Item Health Survey (VR-36) is 36-item measure of health-related quality of life including physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It is often summarized into physical functioning components (PCI) and mental functioning components (MCI), and is one of the most widely utilized and valid measures of physical and psychological well-being.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Week 7
  The SUS a 10-item measure, scored on a 5-point Likert scale, that assesses human-computer interaction. A SUS score above 68 is regarded as above average, and a SUS score above 80 is regarded as high and a score above which participants are likely to recommend the product to friends. The SUS generates a subjective evaluation score using a globally accepted scale and to understand if the system in its current form is sufficiently usable.
Client Satisfaction Questionnaire-8 (CSQ-8) | Week 7
  This 8-item scale measures global satisfaction, perceived quality, and effectiveness of the proposed mental health treatment. This scale has been used in mental health and other health centers and has acceptable internal consistency (.83-.93).
Multidimensional Psychological Flexibility Inventory (MPFI) | Week 7, 3-Month Follow-Up, 6 Month Follow-Up
  A 60-item self-report measure that assesses psychological flexibility, the main mechanism of change proposed in our theoretical model. The MPFI is conceptually grounded in the ACT Hexaflex model, and assesses six dimensions of flexibility (i.e., present moment awareness, self as context, acceptance, contact with values, committed action, cognitive defusion), six dimensions of inflexibility (cognitive fusion, self as context, inaction, lack of contact with values, lack of contact with the present moment, experiential avoidance), and 2 global composite dimensions. The MFPI is sensitive to clinical change and the scales have demonstrated excellent internal consistencies across several subpopulations.
Chronic Pain Acceptance Questionnaire (CPAQ) | Week 7, 3-Month Follow-Up, 6 Month Follow-Up
  A 20-item survey measuring recognition of pain as not negating the ability to live valued life. Pain willingness reflects a pattern of refraining from attempts to control or avoid pain. Higher CPAQ scores indicate higher activity engagement, pain willingness, and overall pain acceptance. The CPAQ is a well-validated measure with high internal consistency and test-retest reliability.
Chronic Pain Values Inventory (CPVI) | Week 7, 3-Month Follow-Up, 6 Month Follow-Up
  A 12-item self-report measure of the extent to which the patient is living in accordance with their values in areas such as work, health, and family, which is related to lower perceived disability and pain-related anxiety, as well as greater reported patient functioning even in the context of high levels of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Erin D. Reilly, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (3):
- United States (3):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reilly ED, Grigorian HL, Heapy AA, Etingen B, Kelly MM, Wolkowicz NR, Girouard CM, Hogan TP, Bernice K, Bickmore T. Assessment of Two Online Interventions for Veterans With Chronic Pain: Protocol for a Randomized Controlled Efficacy Trial. JMIR Res Protoc. 2025 Aug 13;14:e70601. doi: 10.2196/70601. PMID 40802968